CLINICAL TRIAL: NCT00469586
Title: Efficacy and Safety of Inhaled Prandial Insulin Compared to Metformin Plus Glimepiride in Type 2 Diabetes
Brief Title: Efficacy and Safety of Inhaled Insulin Compared to Metformin and Glimepiride in Type 2 Diabetes
Acronym: iINHALE 7
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1998-1787; 2006-004623-12 (EudraCT Number)
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: inhaled human insulin
- B (Experimental)
  Interventions: Drug: inhaled human insulin
- C (Active Comparator)
  Interventions: Drug: metformin; Drug: glimepiride

INTERVENTIONS:
Drug: inhaled human insulin — Treat-to-target dose titration scheme, pre-prandial, inhalation.
  Other Names: NN1998
  Arms: A
Drug: metformin — Tablets, 2000 mg/day.
  Arms: C
Drug: glimepiride — Tablets, 4 mg/day.
  Arms: C
Drug: inhaled human insulin — Treat-to-target dose titration scheme, post-prandial, inhalation.
  Other Names: NN1998
  Arms: B

SUMMARY:
This trial is conducted in Europe, Asia, North America and South America. The aim of this research trial is to compare the efficacy of inhaled insulin to glimepiride and metformin combination therapy in treatment of subjects with type 2 diabetes and to verify the safety of use (hypoglycaemia, pulmonary function, body weight, insulin antibodies and side effects).

DETAILED DESCRIPTION:
The decision to discontinue the development of AERx® is not due to any safety concerns. An analysis concluded that fast-acting inhaled insulin in the form it is known today, is unlikely to offer significant clinical or convenience benefits over injections of modern insulin with pen devices.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treated with OADs for more than or equal to 3 months
* HbA1c greater than or equal to 8.0% and less than or equal to 11.0%
* Body Mass Index (BMI) less than or equal to 40.0 kg/m2

Exclusion Criteria:

* Recurrent major hypoglycaemia
* Current smoking or smoking within the last 6 months
* Impaired hepatic or renal function
* Cardiac problems
* Uncontrolled hypertension
* Proliferative retinopathy or maculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2007-04-26 (Actual); Primary Completion 2008-04-24 (Actual); Study Completion 2008-04-24 (Actual)

PRIMARY OUTCOMES:
HbA1c change from baseline | After 18 weeks of treatment

SECONDARY OUTCOMES:
Adverse events | For the duration of the trial
Body weight | after 18 weeks of treatment
Lung function | after 18 weeks of treatment
Blood glucose | after 18 weeks of treatment
Hypoglycaemia | after 18 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (52):
- Argentina (3):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Mendoza
- Austria (4):
  - Novo Nordisk Investigational Site, Ebreichsdorf
  - Novo Nordisk Investigational Site, Kittsee
  - Novo Nordisk Investigational Site, Salzburg
  - Novo Nordisk Investigational Site, Vienna
- Belgium (6):
  - Novo Nordisk Investigational Site, Arlon
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Borsbeek
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Huy
  - Novo Nordisk Investigational Site, Leuven
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Canada (11):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
  - Novo Nordisk Investigational Site, Mississauga
  - Novo Nordisk Investigational Site, Oshawa
  - Novo Nordisk Investigational Site, Saskatoon
  - Novo Nordisk Investigational Site, Trois-Rivières
- France (6):
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Roubaix
- India (5):
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Bangalore
  - Novo Nordisk Investigational Site, Coimbatore
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Thriruvananthapuram
- Israel (3):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
- Mexico (4):
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
  - Novo Nordisk Investigational Site, Guadalajara
  - Novo Nordisk Investigational Site, Mexico City
- Poland (7):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Mazowieckie
  - Novo Nordisk Investigational Site, Rawa Mazowiecka
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Konya

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com